CLINICAL TRIAL: NCT07193654
Title: Stupp Regimen Combined With Intrathecal Injection of Thiotepa for the Treatment of Glioblastoma With Ventricular Invasion or Meningeal Metastasis：a Prospective, Single-Arm, Exploratory Study
Brief Title: Stupp Treatment With Intrathecal Injection of Thiotepa for Glioblastoma With Advanced Spread
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y2025-0127
Record Dates: First submitted 2025-03-24; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma (GBM)
Keywords: brain ventricles invasion; meningeal metastasis; Intrathecal chemotherapy
MeSH Terms: conditions — Glioblastoma; Meningeal Carcinomatosis | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stupp plus intrathecal injection of thiotepa (Experimental)
  Interventions: Drug: Intrathecal injection of thiotepa; Drug: Stupp regimen (oral temozolomide); Radiation: Radical radiotherapy; Procedure: Maximal surgical resection

INTERVENTIONS:
Drug: Intrathecal injection of thiotepa — Intrathecal injection of thiotepa: Administered via lumbar puncture or OMMAYA reservoir according to the study protocol.
Drug: Stupp regimen (oral temozolomide) — Stupp regimen (oral temozolomide)::75 mg/m² daily during radiotherapy; 150-200 mg/m² daily for 5 days every 28 days for 6 cycles after radiotherapy;
Radiation: Radical radiotherapy — Radical radiotherapy: Delivery of 60 Gy of radiation, typically divided into 30 fractions of 2 Gy each;
Procedure: Maximal surgical resection — Maximal surgical resection: Removal of as much tumor as possible while preserving neurological function;

SUMMARY:
The goal of this clinical trial is to learn if a combined treatment approach can treat glioblastoma (GBM) with ventricular invasion or meningeal metastasis in adults. The main questions it aims to answer are:

Does the combined treatment of radical radiotherapy, the Stupp regimen (oral temozolomide), and intrathecal injection of thiotepa improve progression-free survival compared to standard treatment alone?

Does the combined treatment improve overall survival compared to standard treatment alone?

Participants will:

* Undergo maximal surgical resection of the tumor；
* Receive radical radiotherapy；
* Take oral temozolomide according to the Stupp regimen；
* Receive intrathecal injections of thiotepa。

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common and aggressive primary malignant brain tumor in adults, with a dismal prognosis despite standard treatment. The standard treatment for GBM, which includes surgery, radiotherapy, and chemotherapy with temozolomide (known as the Stupp regimen), has remained largely unchanged for over two decades. Patients with GBM who have tumor invasion of the brain ventricles or meningeal metastasis face an even worse prognosis, with significantly shorter progression-free survival and overall survival compared to patients without these complications. The blood-brain barrier poses a significant challenge to effective chemotherapy delivery, limiting the efficacy of systemic treatments for central nervous system tumors. Intrathecal chemotherapy administration represents a promising strategy to overcome this barrier by directly delivering chemotherapeutic agents into the cerebrospinal fluid, potentially improving tumor control and survival outcomes in patients at high risk for intraventricular dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 75, any gender.
* Newly diagnosed WHO grade 4 brain tumor with at least one evaluable lesion, imaging suggesting ventricular or meningeal invasion.
* History of intraoperative intraventricular or cisternal opening.
* Malignant cells found in cerebrospinal fluid pre-radiotherapy.
* ECOG score 0 - 2, expected survival≥3 months.
* Stable neurological symptoms for over 7 days.
* Neutrophil count≥1.5×10⁹/L, hemoglobin≥90 g/L, platelet count≥75×10⁹/L.
* PT/INR and PTT≤1.5×upper limit of normal.
* Total bilirubin≤1.5×upper limit of normal, AST and ALT≤1.5×upper limit of normal, albumin≥30 g/L, creatinine≤2×upper limit of normal, calculated or 24-hour urine creatinine clearance rate≥50 mL/min.
* Agree to effective contraception from first to 3 months after last dose.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Active infection within 7 days before starting study drug requiring IV antibiotics or therapeutic warfarin.
* Other malignancies in past 5 years.
* HIV/AIDS history; past immunodeficiency, or active autoimmune disease needing systemic treatment.
* Severe medical, neurological, or psychiatric conditions preventing full adherence to study treatment or assessments.
* Ventricular drainage tube rupture or inability to undergo lumbar puncture.
* Uncontrolled chronic diseases like diabetes, CHF, liver cirrhosis, or CKD.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety assessment | From first dose of study treatment until 30 days after last dose, assessed up to 52 weeks.
  Incidence and severity of treatment-related adverse events using CTCAE 5.0.

SECONDARY OUTCOMES:
Progression-free survival | 3 months,6 months and 1 year after treatment
  Time from treatment initiation until disease progression( RECIST1.1 )
Overall survival | Until date of death from any cause, assessed up to 24 months.
  Time from treatment initiation until death

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Hangzhou, Zhejiang, China